CLINICAL TRIAL: NCT00224601
Title: Early Detection of Pre-cancer Lesions in Adults With Hereditary Nonpolyposis Colorectal Cancer (HNPCC) Syndrome: Assessment of Coloscopy With Chromoscopy Benefit
Brief Title: CHROENDOHNPCC: Early Detection of Pre-cancer Lesions in Adults With Hereditary Nonpolyposis Colorectal Cancer Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha DJANE, Department of Clinical Research of developpement
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P040423
Record Dates: First submitted 2005-09-16; First posted 2005-09-23 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-07

CONDITIONS: Colorectal Neoplasms, Hereditary Nonpolyposis
Keywords: Colorectal cancer; HNPCC; Diagnosis; Coloscopy; Chromoscopy; Indigo carmine; Colorectal Neoplasms; Hereditary Nonpolyposis
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Disease | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Colonoscopy with chromoscopy

SUMMARY:
The aim of the study is to test the hypothesis that a chromoscopy colonoscopy is able to increase by 50 % the number of pre-cancer lesions or early cancer detected in patients with HNPCC syndrome, compared to a routine colonoscopy without chromoscopy.

DETAILED DESCRIPTION:
Patient with HNPCC syndrome confirmed by a mutation (MLH1, MSH2, MHS1) are involved in the study. Patient have 2 colonoscopy back to back. The second coloscopy is associated to chromoscopy with carmin indigo. Endoscopist are randomised for the colonoscopy with chromoscopy and are un-awarded of the result of the first colonoscopy. Histopathology of the polyp are noted. The follow up were 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MLH1, MSH2 or MSH6 mutation.
* Patients concerned by early detection colonoscopy.

Exclusion Criteria:

* Coloscopy of tracking since less 1an
* occlusive Syndrome contra-indicating the preparation for a total coloscopies
* Colectomies
* medical Conditions or serious illnesses contra-indicating a coloscopy of screening
* pregnant Woman or nursing
* Anomaly of coagulation contra-indicating the realization of biopsies and/or the exeresis of the lesion colorectal

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of pre-cancer lesions or early cancer detected. | during the procedure

SECONDARY OUTCOMES:
Anatomopathologic criteria (size of lesions, …). | during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CELLIER, Pr,MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Mention JJ, Ben Ahmed M, Begue B, Barbe U, Verkarre V, Asnafi V, Colombel JF, Cugnenc PH, Ruemmele FM, McIntyre E, Brousse N, Cellier C, Cerf-Bensussan N. Interleukin 15: a key to disrupted intraepithelial lymphocyte homeostasis and lymphomagenesis in celiac disease. Gastroenterology. 2003 Sep;125(3):730-45. doi: 10.1016/s0016-5085(03)01047-3. PMID 12949719